CLINICAL TRIAL: NCT03767868
Title: A Different Indicator of Successful Peripheral Nerve Block
Brief Title: An Indicator of Successful Peripheral Nerve Block
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH27
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2018-12

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: color change in nail polish — The determination of color change in nail polish will be based on differences in skin temperature before and after the block.

SUMMARY:
The aim of the study was to investigate whether a color changing nail polish would be an indicator to assess infraclavicular brachial plexus block success based on skin temperature differences before and after performed the block.

DETAILED DESCRIPTION:
After performed the block, sensory and motor block assessments will be carried out by blinded observer every 5 min after needle removal for 30 min in the regions of the radial, median, ulnar, and musculocutaneous nerves of the forearm. Skin temperature measurements will be performed from both the anesthetized side and the contralateral arm before the procedure and every 5 min for 30 min by a blinded observer. Before the block, the color changing nail polish will be applied to all hand nails of the patient. An independent observer will photograph the reaction of the nail polish (i.e. color change) in both hands immediately after application of nail polish and at two minute intervals for 30 min after performing the block. Two blinded observers were reviewed the digital photographs. They were asked to compare the colors of nail polish in both hands and to score the difference based on a three-point scale (0: absolutely no difference, 1: I am not sure, 2: indisputable difference)

ELIGIBILITY:
Inclusion Criteria:

* patients who received infraclavicular brachial plexus block for elective elbow, forearm, wrist, or hand surgery
* American Society of Anesthesiologists class I, II or III

Exclusion Criteria:

* patients <18 years old
* >65 years old
* body mass index (BMI) <20 or >35 kg/m2
* inability to provide written informed consent
* refusal of regional anesthesia
* pregnancy
* contraindication for regional anesthesia
* peripheral neurological disease,
* Raynaud disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between 18 and 65 years of age with infraclavicular brachial lexus block for elective elbow, forearm, wrist, or hand surgery , were selected in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Differences in the color of nail polish | 30 minutes
  The photographs showing if there is the reaction of color of nail polish will be assessed after study completion by independent observers. They will be asked to compare the colors of nail polish before and after block performance in both hands and to rate the difference based on a three-point scale (0: absolutely no difference, 1: I am not sure, 2: indisputable difference).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, MD, Study Director — Antalya Training and Research Hospital; Ulku Arslan, MD, Principal Investigator — Karabuk University; Ferhat Enginar, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Kavakli AS, Enginar F, Arslan U, Ozdemir F. Thermochromic nail polish as a novel indicator to predict infraclavicular brachial plexus block success: A prospective cohort study. Eur J Anaesthesiol. 2019 Dec;36(12):911-917. doi: 10.1097/EJA.0000000000001091. PMID 31592901